CLINICAL TRIAL: NCT04679324
Title: The Role of Mucosal Microbiome in the Development, Clearance and Recurrence of Clostridiodes Difficile Infection
Brief Title: The Role of Mucosal Microbiome in the Development, Clearance and Recurrence of Clostridioides Difficile Infection
Status: Withdrawn | Type: Observational
Why Stopped: C. difficile symptoms preclude participants from attending research study visits.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005222
Record Dates: First submitted 2020-12-09; First posted 2020-12-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sigmoid colon biopsies, stool samples, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is being done to identify types of bacteria associated with the lining of the large intestine in people who have recently been diagnosed with C. difficile infection to determine if there are features associated with development, clearance, and recurrence of disease.

DETAILED DESCRIPTION:
Patients who were recently diagnosed with C. difficile infection will undergo assessment of both before treatment and after completing treatment to study the presence of C. difficile in the colonic mucosa pre as well as assessment for microbiome and patient/clinical factors that may contribute to disease recurrence. Assessment will include sigmoid colon biopsies, blood draw, stool samples and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Confirmed C. difficile infection based on positive C. difficile toxin PCR testing and clinical evidence of diarrhea

Exclusion Criteria:

* Known active pregnancy
* Prior diagnosis of C. difficile infection within 2 months of this diagnosis
* Other known active gastrointestinal infectious process
* Vulnerable adults
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recently diagnosed with C. difficile infection (not defined as recurrent) without underlying inflammatory GI conditions
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Disease recurrence | 8 weeks post treatment of C.difficile infection
  Based on clinical stool testing and symptoms

SECONDARY OUTCOMES:
Change in mucosal presence of C. difficile | Baseline, approximately 1-14 days post treatment of C. difficile infection
  Identification of C. difficile within the colonic mucosa on stained slides from sigmoid biopsy samples

CONTACTS AND LOCATIONS:
Overall Officials: Purna Kashyap, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials